CLINICAL TRIAL: NCT06835205
Title: Prevention Workshop to Address Bullying Behaviors in Schools: A Cluster Randomized Controlled Trial
Brief Title: Prevention Workshop to Address Bullying Behaviors in Schools
Acronym: APACHES
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Université Lumière Lyon 2 (Other); University Grenoble Alps (Other); Maison des Sciences de l'Homme et de la société (Unknown); Grenoble Academy (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PREPS-22-0015
Record Dates: First submitted 2025-01-13; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Bullying of Child; Child Behavior Disorders; Social Behavior; Mental Health; Interpersonal Relations; School Health Services; Prevention and Control
Keywords: Bullying Prevention; Psychosocial Skills; Elementary Education; Health Education; Student Well-Being; Cluster Randomized Trial; TEAL Program; School Climate; Public Health Intervention
MeSH Terms: conditions — Child Behavior Disorders; Social Behavior; Psychological Well-Being; Health Education

STUDY DESIGN:
Intervention Model Description: This is a cluster randomized controlled trial where classrooms are randomized into two groups: the intervention group receives the TEAL program, and the control group participates in unrelated health education sessions.
Masking Description: Although the study is open-label for participants, care providers, and investigators, the statistician conducting the data analysis will remain blinded to group allocation. This ensures unbiased interpretation of the results.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (TEAL Program) (Experimental): Students in this group will receive the "Tous Épanouis à l'École" (TEAL) program, a five-session intervention aimed at developing psychosocial skills, including empathy, communication, and social proximity. Sessions will be conducted by trained healthcare students as part of their Service Sanitaire curriculum. The program focuses on reducing bullying behaviors and improving classroom climate.
  Interventions: Behavioral: Tous Épanouis à l'École (TEAL Program)
- Control Group (Standard Health Education) (Active Comparator): Students in this group will participate in five health education sessions on topics unrelated to bullying (e.g., nutrition, sleep hygiene). These sessions will also be delivered by healthcare students following the standard Service Sanitaire training curriculum.
  Interventions: Behavioral: Standard Health Education Sessions

INTERVENTIONS:
Behavioral: Tous Épanouis à l'École (TEAL Program) — The TEAL Program is a structured, five-session behavioral intervention targeting psychosocial skill development in children. Delivered by healthcare students in elementary school classrooms, the program includes interactive activities designed to improve communication, empathy, social proximity, and prosocial behaviors. The intervention aims to reduce bullying behaviors (victims and aggressors) and enhance classroom climate. Each session is guided by a detailed manual and includes active participation from students and their teachers.
  Arms: Intervention Group (TEAL Program)
Behavioral: Standard Health Education Sessions — This intervention consists of five sessions on general health topics unrelated to bullying, such as nutrition, sleep hygiene, and physical activity. The sessions are facilitated by healthcare students as part of their Service Sanitaire training. These sessions provide a comparable structure and duration to the TEAL program but do not address bullying prevention.
  Arms: Control Group (Standard Health Education)

SUMMARY:
This study, titled APACHES, is a cluster randomized controlled trial aimed at evaluating the effectiveness of a school-based prevention program, "Tous Épanouis à l'École" (TEAL), conducted by healthcare students as part of their mandatory public health service curriculum. The TEAL program consists of five interactive sessions focused on developing psychosocial skills (e.g., communication, empathy, collaboration) among elementary school students (grades CE2-CM1-CM2) in the Grenoble Academy. The primary objective is to assess whether the program reduces the prevalence of bullying behaviors (victims and/or aggressors) compared to standard preventive actions on unrelated themes. The study involves 36 classrooms across 18 schools, with data collected at three time points: before, one month after, and four months after the intervention. Secondary objectives include evaluating social proximity, altruistic behaviors, and qualitative perceptions from students, teachers, and facilitators.

DETAILED DESCRIPTION:
Bullying is a critical public health issue with severe consequences for children's psychological development, academic success, and long-term health outcomes. The APACHES study evaluates the effectiveness of the TEAL program, a psychosocial skills training intervention tailored to reduce bullying behaviors and improve classroom climate. The intervention will be delivered by healthcare students (from medicine, midwifery, pharmacy, and nursing) as part of their Service Sanitaire curriculum.

The study follows a pragmatic design with a cluster randomized controlled methodology. Classrooms in participating schools are randomized into two groups: an intervention group receiving the TEAL program and a control group undergoing alternative health education sessions. The TEAL program is structured around active and participatory learning, including sessions on emotional awareness, communication, empathy, and collective problem-solving. A total of 900 students from 36 classrooms (approximately 450 per group) will participate.

Objectives Primary Objective: To determine whether the TEAL program reduces the prevalence of bullying (victims and/or aggressors) by comparing baseline and follow-up outcomes.

Secondary Objectives: To explore improvements in social proximity, altruistic behaviors, and psychosocial skills; to collect qualitative feedback from students, facilitators, and teachers about the intervention.

Data Collection and Outcomes Quantitative data will be collected using validated questionnaires (e.g., Revised Bully/Victim Questionnaire) administered at three time points: pre-intervention (T1), one month post-intervention (T2), and four months post-intervention (T3). Secondary outcomes, including social proximity and altruism, will also be assessed. Qualitative data will be gathered through interviews and focus groups to evaluate participants' experiences and perceptions.

Significance This study aims to address a pressing public health need by leveraging healthcare students' involvement in primary prevention. If effective, the TEAL program could be scaled nationally across France, contributing to the broader goal of improving psychosocial environments in schools and mitigating the long-term effects of bullying.

ELIGIBILITY:
Inclusion Criteria:

* Students enrolled in grades CE2, CM1, or CM2 in participating schools.
* Parents or legal guardians have provided signed informed consent for their child to participate in the study.
* The child is available to attend all scheduled intervention sessions.

Exclusion Criteria:

* Students whose parents or legal guardians have not provided signed informed consent.
* Students with medical or behavioral conditions that might prevent full participation in the sessions (e.g., requiring additional support not available during the study).
* Students not attending the school on a regular basis.

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 900 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Bullying Behaviors (Victims and/or Aggressors) | Change from baseline (T1) to one month after the intervention (T2).
  The proportion of students identified as victims, aggressors, or victim-aggressors based on the Revised Bully/Victim Questionnaire (rBVQ). Measured at three time points: before the intervention (T1), one month after the intervention (T2), and four months after the intervention (T3).

SECONDARY OUTCOMES:
Change in Social Proximity Score | Change from baseline (T1) to one month after the intervention (T2).
  Assessment of the social proximity among students using a validated scale. The change in scores will be measured at T1, T2, and T3 to evaluate the intervention's impact on fostering closer social relationships.
Change in Psychosocial Skills | Change from baseline (T1) to one month after the intervention (T2).
  Improvement in psychosocial skills such as empathy, communication, and emotional regulation, measured via a validated psychosocial skill scale. Changes are assessed at T1, T2, and T3.
Change in Altruistic Behaviors | Change from baseline (T1) to one month after the intervention (T2).
  Improvement in students' altruistic behaviors, assessed using the French version of the Child Altruism Scale (20 items). Measurements occur at T1, T2, and T3.
Perception of the Intervention by Healthcare Students (Focus Groups) | Collected one month after the intervention (T2)
  Exploration of the perceptions and experiences of healthcare students who facilitated the TEAL program, gathered through focus groups. Topics include perceived impact, challenges, and learning outcomes from the intervention.
Perception of the Intervention by Elementary School Teachers (Interviews) | Collected one month after the intervention (T2)
  Feedback from teachers in the TEAL group on the program's impact on classroom dynamics, bullying behaviors, and overall implementation. Data are collected through semi-structured interviews.
Perception of the Intervention by Students (Interviews) | Collected one month after the intervention (T2)
  Qualitative feedback from children in the TEAL group on their experiences with the program, including perceived benefits, engagement, and understanding of key themes. Data are collected via semi-structured interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Bastien Boussat, MD, PhD, Principal Investigator — University Grenoble Alpes, Faculty of Medicine
Locations (1):
- Académie de Grenoble, Grenoble, France

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie the results reported in the publication (after de-identification) will be shared with researchers upon reasonable request. Data will include:
  Demographic variables Outcome measures (e.g., bullying behaviors, psychosocial skills, and social proximity scores) Qualitative data (e.g., thematic analysis results from focus groups and interviews) Data will be available beginning 6 months after publication and ending 5 years after publication. Requests for data sharing must include a detailed proposal that is approved by the study's steering committee. Access will be granted through a secure data-sharing platform. Contact information for data requests: bboussat@chu-grenoble.fr.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD and supporting information will be available starting 6 months after publication of the primary results. Data and documents will remain accessible for 5 years post-publication.
Access Criteria: Researchers with a scientifically sound proposal may request access to the IPD and supporting documents.
  Requests must include a detailed research plan and intended use of the data, subject to approval by the study's steering committee.
  Approved users will sign a data access agreement and will access the data through a secure data-sharing platform.
  Contact: bboussat@chu-grenoble.fr.